CLINICAL TRIAL: NCT03735810
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Single and Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of LBS-008 in Healthy Adult Subjects
Brief Title: Safety and Tolerability Study of LBS-008 in Healthy Adult Subjects After Single and Multiple Doses
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: RBP4 Pty Ltd (Industry)
Collaborators: Belite Bio, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: LBS-008-CT01
Record Dates: First submitted 2018-11-07; First posted 2018-11-08 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2019-08

CONDITIONS: Healthy Volunteer

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (9):
- SAD - Cohort 1 (Experimental): 50 mg LBS-008 or placebo
  Interventions: Drug: LBS-008; Drug: Placebos
- SAD - Cohort 2 (Experimental): 100 mg LBS-008 or placebo
  Interventions: Drug: LBS-008; Drug: Placebos
- SAD - Cohort 3 (Experimental): 200 mg LBS-008 or placebo
  Interventions: Drug: LBS-008; Drug: Placebos
- SAD - Cohort 4 (Experimental): 400 mg LBS-008 or placebo
  Interventions: Drug: LBS-008; Drug: Placebos
- SAD - Cohort 5 (Experimental): 25 mg LBS-008 or placebo
  Interventions: Drug: LBS-008; Drug: Placebos
- MAD - Cohort 1 (Experimental): 10 mg LBS-008 or placebo
  Interventions: Drug: LBS-008; Drug: Placebos
- MAD - Cohort 2 (Experimental): 25 mg LBS-008 or placebo
  Interventions: Drug: LBS-008; Drug: Placebos
- MAD - Cohort 3 (Experimental): 5 mg LBS-008 or placebo
  Interventions: Drug: LBS-008; Drug: Placebos
- MAD - Cohort 4 (Experimental): 12 mg LBS-008 or placebo
  Interventions: Drug: LBS-008; Drug: Placebos

INTERVENTIONS:
Drug: LBS-008 — LBS-008 oral capsules
Drug: Placebos — Oral capsules

SUMMARY:
This is a single center, randomized, double-blind, placebo-controlled, Single Ascending Dose (SAD) and Multiple Ascending Dose (MAD) study is planned to assess safety, pharmacokinetics (PK), and pharmacodynamics of LBS-008 in healthy adult volunteers.

ELIGIBILITY:
Inclusion Criteria:

* The subject is male or female, 18 to 65 years of age, inclusive, at screening.
* The subject voluntarily consents to participate in this study and provides written informed consent before the start of any study-specific procedures.
* The subject is willing and able to remain in the study unit for the entire duration of the confinement period and return for outpatient visits.
* Female subjects must be of nonchildbearing potential (defined as surgically sterile [i.e., had a bilateral tubal ligation, hysterectomy, or bilateral oophorectomy at least 6 months before the dose of study drug] or postmenopausal for at least 1 year before study drug administration confirmed by FSH test at screening; FSH level >40 mIU/mL). Female subjects may also be considered of non-childbearing if they have a confirmed medical condition which would deem the subject as infertile. E.g. MRKH Syndrome (Mullerian Agenesis) or another applicable condition.
* Male subjects must be surgically sterile (i.e., vasectomy) for at least 3 months before screening; or remain abstinent or agree to use a highly effective form of contraception when sexually active with a female partner for 90 days after study drug administration. Highly effective contraception requires use of a condom and appropriate contraceptive measures for your female partner (i.e. oral, injected or implanted hormonal methods, or placement of an intrauterine device or intrauterine system). This requirement does not apply to subjects in a same sex relationship and female partners of non-childbearing potential.
* The subject has a body mass index (BMI) of 18 to 30 kg/m2, inclusive, and weighs 50 to 100 kg (110 to 220 pounds), inclusive, at screening and check-in.
* The subject is considered to be in stable health by the investigator.
* The subject agrees to comply with all protocol requirements.

Exclusion Criteria:

* Any significant acute or chronic medical illness including history or presence of clinically significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, oncologic, or psychiatric disease
* Vitamin A deficiency.
* Any recent viral or bacterial infection.
* Participated in any clinical study in last 6 weeks.
* History of significant drug allergy
* History of significant vision, ocular or retinal disorder.
* Recent surgery, blood transfusion, drug or alcohol abuse and use of tobacco or nicotine containing products in past month.
* Evidence of organ dysfunction or any clinically significant deviation from normal in physical examination, vital signs, ECGs, or clinical laboratory determinations Other protocol-defined inclusion/exclusion criteria could apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2018-11-15 (Actual); Primary Completion 2019-09-16 (Actual); Study Completion 2019-09-16 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve from time 0 to the last timepoint with quantifiable concentration (AUC0-t) | SAD portion: Day 1 to Day 8; MAD portion: Day 1 to Day 28
Area under the plasma concentration versus time curve from time 0 extrapolated to infinity (AUC0-inf) | SAD portion: Day 1 to Day 8; MAD portion: Day 1 to Day 28
Maximum observed plasma concentration (Cmax) | SAD portion: Day 1 to Day 6; MAD portion: Day 1 to Day 28
Time to maximum observed plasma concentration (Tmax) | SAD portion: Day 1 to Day 8; MAD portion: Day 1 to Day 28
Terminal elimination rate constant | SAD portion: Day 1 to Day 8; MAD portion: Day 1 to Day 28
Terminal phase half-life (t1/2) | SAD portion: Day 1 to Day 8; MAD portion: Day 1 to Day 28
Apparent total body clearance (CL/F) | SAD portion: Day 1 to Day 8; MAD portion: Day 1 to Day 28
Apparent volume of distribution (Vz/F) | SAD portion: Day 1 to Day 8; MAD portion: Day 1 to Day 28
Number of participants with Adverse Events (AEs), Serious Adverse Events (SAEs) and AEs leading to discontinuation. | SAD portion: Day 1 to Day 8; MAD portion: Day 1 to Day 28

CONTACTS AND LOCATIONS:
Locations (1):
- Linear Clinical Research, Perth, Australia

IPD SHARING:
Plan to Share IPD: No
After completion of the study, data may be considered for reporting at a scientific meeting or for publication in a scientific journal. In these cases, the sponsor will be responsible for these activities and will work with the investigators to determine how the manuscript is written and edited, the number and order of authors, the publication to which it will be submitted, and any other related issues. The sponsor has final approval authority of all such issues. Data are the property of the sponsor and cannot be published without their prior authorization, but data and any publication thereof will not be unduly withheld.